CLINICAL TRIAL: NCT03021356
Title: Prospective Randomized Comparison of TrIfecta and Perimount Magna Ease
Brief Title: Comparison of TrIfecta and Perimount Magna Ease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kerckhoff Klinik (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COTRIP
Record Dates: First submitted 2017-01-08; First posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Aortic Xenograft Hemodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trifecta aortic xenograft (Active Comparator): The Trifecta aortic xenograft is implanted in these patients.
  Interventions: Device: Aortic xenograft
- Magna Ease aortic xenograft (Active Comparator): The Magna Ease aortic xenograft is implanted in these patients.
  Interventions: Device: Aortic xenograft

INTERVENTIONS:
Device: Aortic xenograft — After randomization, the aortic xenograft is implanted in the standard fashion

SUMMARY:
The hemodynamic performance of two supraannular aortic xenografts (Trifecta, St. Jude Medical and Perimount Magna Ease, Edwards Lifescience) will be compared using rest- and stress echocardiography in a randomized prospective study. Furthermore, the prostheses' influence on postoperative outcome will be compared using spiroergometry, quality of life questionnaire and heart failure biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 75 years
* Elective aortic valve replacement in patients with predominant aortic stenosis

  * including concomitant CABG and/or atrial fibrillation ablation and/or supracoronary aortic replacement
* Informed consent including willingness for stress echocardiography, spiroergometry and quality of life examination after 6 months.
* Native German speakers (quality of life questionnaire in German language)

Exclusion Criteria:

* Isolated aortic regurgitation
* Concomitant aortic regurgitation > 2°
* Endocarditis
* LVEF <40%
* Concomitant other valve surgery
* s/p valve surgery
* Contraindication for stress echocardiography

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Transprosthetic pressure gradient at stress exercise echocardiography | Echo at follow up stress echo (at 10 months)

SECONDARY OUTCOMES:
Transprosthetic pressure gradient at discharge echo | Echo at discharge (usually postoperative day 5 to 7)
Left ventricular mass regression calculated by echocardiography (gram) | Echo at discharge and at follow up (usually at postoperative day 5 to 7 and at 10 months)
Quality of life using the EQ-5D-3L questionnaire | 1 to 5 days before surgery and at follow up (10 months)
BNP plasma level | 1 to 5 days before surgery and at follow up (10 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Kerckhoff Klinik, Bad Nauheim, Germany

IPD SHARING:
Plan to Share IPD: No